CLINICAL TRIAL: NCT07204171
Title: Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of Oral MG001
Brief Title: Phase 1 Study of Oral MG001
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Altasciences Clinical Kansas, Inc. (Unknown); Technical Resources International, Inc. (TRI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-MG001-Ph1a-001; 75N95023D20019 (Other: National Institute on Drug Abuse (NIDA))
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Safety and Tolerability in Healthy Subjects
Keywords: mitragynine; kratom; opioid use disorder; opioid withdrawal
MeSH Terms: conditions — Opioid-Related Disorders | interventions — mitragynine

STUDY DESIGN:
Intervention Model Description: This is first-in-human (FIH), randomized, double-blind, placebo-controlled, single ascending dose (SAD), phase I study in healthy participants. Four single ascending dose levels under fasting conditions are proposed.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 25 mg dose (Experimental): oral administration in fasted state
  Interventions: Drug: mitragynine
- 50 mg dose (Experimental): oral administration in fasted state
  Interventions: Drug: mitragynine
- 75 mg dose (Experimental): oral administration in fasted state
  Interventions: Drug: mitragynine
- 100 mg dose (Experimental): oral administration in fasted state
  Interventions: Drug: mitragynine
- Placebo (Placebo Comparator): oral administration in fasted state
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mitragynine — Mu opioid receptor partial agonist
  Arms: 100 mg dose; 25 mg dose; 50 mg dose; 75 mg dose
Drug: Placebo — Each of the four dose groups of n=8 participants will be assigned to active drug or placebo in the ration 6:2.
  Arms: Placebo

SUMMARY:
This research study is the first time the new medication MG001 is being tested in people. MG001 is a formulation of mitragynine, a compound that comes from a plant called Mitragyna speciosa (sometimes known as kratom), which some people use on their own to help manage symptoms of opioid withdrawal. The purpose of this study is to understand how safe MG001 is, how well it is tolerated, and how the body processes it. About 32 healthy adult volunteers, both men and women, will take part. Before joining, participants will undergo screening tests up to four weeks in advance to make sure they are eligible and healthy enough. On the day before dosing, participants will be admitted to the clinic for final health checks, and those who qualify will be randomly assigned-by chance, like flipping a coin-to receive either a single dose of MG001 or a placebo (an inactive substance). Neither the participants nor the staff giving the medicine will know which one is given. The study drug will be administered after at least 10 hours of fasting, and participants will then remain in the research clinic under close medical observation for three nights, until Day 4. During this time, doctors and nurses will monitor participants' health, look for any side effects, and collect blood samples to see how MG001 moves through the body. A follow-up clinic visit on Day 7 will provide one last check-in and blood test. This design helps researchers gather important first information on the safety and tolerability of MG001, while protecting the health and well-being of participants.

DETAILED DESCRIPTION:
This first in human (FIH), randomized, double-blind, placebo-controlled, single ascending dose (SAD) phase I study in healthy participants is designed to assess the safety and tolerability of MG001. Approximately 32 healthy male and female volunteers will be enrolled.

Participants will be screened for eligibility as outpatients and inpatients. Outpatient screening will occur between Day -28 and Day -2. On Study Day -1, participants will undergo the clinic intake to screen for continued eligibility. Once a participant has been determined to be eligible, the participant will be randomized to receive either MG001 or placebo. Participants will receive the assigned treatment on Day 1 after participants have fasted for at least 10 hours. Safety and PK assessments will start on Day 1 and continue until discharge.

Participants will be discharged from the research clinic on Day 4 and seen for a follow-up visit on Day 7 , when the last PK sample will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male or female volunteer between 18 and 65 years of age, inclusive, at the time of consent.
2. Has a body mass index (BMI) within the range of 18.0 to 32.0 kg/m2 and a minimum weight of at least 50.0 kg at screening.
3. Has a recent history of oral opioid use , defined as using prescription or recreational oral opioids at least once during the 30-day period preceding screening.
4. Is able to speak English sufficiently to understand the study procedures and provide written informed consent to participate in the study.
5. Has no clinically significant concurrent medical conditions determined by medical history, physical examination, clinical laboratory test , vital signs, and 12-lead ECG.
6. A female study participant must be of non-childbearing potential - should be surgically sterile (i.e., has undergone complete hysterectomy, bilateral oophorectomy, bilateral salpingectomy or tubal ligation/occlusion) or in a menopausal state (at least 1 year without menses), as confirmed by follicle stimulating hormone (FSH) levels (≥40 mIU/mL).

   If a male study participant that engages in sexual activity that has the risk of pregnancy, must agree to use a double barrier method (e.g., condom and spermicide) and agree to not donate sperm during the study and for at least 90 days after the last dose of the study medication.
7. Is able and willing to comply with protocol requirements and the rules and regulations of the study site and is likely to complete all the study treatments.

Exclusion Criteria:

1. Has any clinically significant finding within one year of Screening on medical history, physical examination, complete neurological examination, clinical laboratory test, vital signs (including hemoglobin saturation assessed by pulse oximetry, RR, HR, BP, oral body temperature ), or ECGs that contraindicate participation in the study. This includes but is not limited to history of or current cardiac, hepatic, renal, neurologic, gastrointestinal (GI) , pulmonary, endocrinologic, hematologic, or immunologic disease or history of malignancy.
2. Has clinically significant psychiatric symptoms and/or psychiatric comorbidities (schizophrenia, bipolar disorders, mania, unipolar depression, disruptive behaviors, etc.), or a history of such within one year of screening. Psychiatric assessment will be conducted by a Qualified Mental Health Professional using the Mini-International Neuropsychiatric Interview (MINI).
3. Has a history of suicide attempts or evidence of suicidal ideation based on the Columbia-Suicide Severity Rating Scale (C-SSRS):

   * Any lifetime history of serious or recurrent suicidal behavior.
   * Previous history of suicidal behaviors in the past 10 years.
   * Suicidal ideation with or without a plan (active or passive, respectively) in the past year.
4. Has a history of epilepsy, seizure disorder, or head trauma with neurological sequelae (e.g., loss of consciousness that required hospitalization); current anorexia nervosa or bulimia; or any other conditions that increase seizure risk in the opinion of the study clinician.
5. Has a history of thyroid and/or parathyroid disease or abnormal T4 or PTH levels.
6. Has evidence of second or third degree heart block, atrial fibrillation, atrial flutter, prolongation of the QTc, or any other finding on the screening ECG that, in the opinion of the study medical clinician, would preclude safe participation in the study.
7. Has any clinically significant abnormal laboratory values
8. Has taken kratom or any investigational drug in another study within 30 days of study consent.
9. Requires treatment with opioid-containing medications (e.g., opioid analgesics) during the study period.
10. Has used opioids intravenously or on 3 or more consecutive days during the 30 day period preceding screening.
11. Has a sitting systolic blood pressure (SBP) >140 mmHg, diastolic BP (DBP) >90 mmHg or HR <50 or >100 beats per minute (BPM) at screening and clinic intake.
12. Has orthostatic hypotension, defined as a 20 mmHg reduction in SBP and 10 mmHg in DBP.
13. Has an O2 saturation, defined as the percentage of hemoglobin in the blood that is carrying oxygen, below 95% from a 10 second reading.
14. Has donated blood (excluding plasma donation) of approximately 500 mL within 56 days prior to screening.
15. Has donated plasma within 7 days prior to screening.
16. Has taken any concomitant medications, including prescription, over-the-counter, dietary supplements, herbal products, vitamins, or medications interacting with CYP3A4, CYP2D6, or CYP1A2 within 14 days or 5-half-lives (whichever is longer) prior to study drug administration, and throughout the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events in Healthy Adult Participants | 4 days in clinic, follow-up on day 7
  The incidence of treatment-emergent adverse events will be measured using a combination of data collection methods, including tracking adverse events and assessing their onset or worsening relative to the initiation of treatment. The most recent version of the Medical Dictionary for Regulatory Activities (MedDRA) preferred terms will be used to classify adverse events, including their relationship to the treatment and maximum severity. Events will be identified either through subject self-report or clinically significant abnormal findings on: (i) Physical examination (ii) Vital signs assessments (heart rate (BPM), blood pressure (mmHg), respiration rate (BPM), hemoglobin saturation (%) and temperature (F)) (iii) ECG assessment (QTcF) as determined by the Investigator/consulting board-certified cardiologist (iv) pupil constriction (mm) (v) sedation as measured by VAS (score) and MOAA/S (score (vi) Clinical Laboratory Assessments

SECONDARY OUTCOMES:
Cmax | 144 hours
  maximum observed plasma concentration (ng/mL)
AUC | 144 hours
  area under the concentration-time curve (mg*h/L)
Tmax | 144 hours
  time of maximum observed plasma concentration (hours)
half-life (t1/2) | 144 hours
  MG001 elimination half-life (hours)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Solarczyk Donnelly, MS, RAC, Study Director — National Institute on Drug Abuse, NIH
Locations (1):
- Altasciences Clinical Kansas, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided